CLINICAL TRIAL: NCT06307730
Title: Duration of Antibiotic Treatment for Infectious Pneumonia in Eldery Subjects
Brief Title: Application of the Recommendations of the SPLIF (French Society of Infectious Pathology) in a Geriatric Population on the Duration of Treatment for Bacterial Pneumonia
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0033_GERIATRIE
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pneumonia, Bacterial; Pneumopathy
Keywords: pneumopathy; Bacterial; nosocomial
MeSH Terms: conditions — Pneumonia, Bacterial; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumopathy is the leading cause of death from infectious disease in the elderly. Prior to 2021, the recommended duration of antibiotic therapy for pneumonia, in adults, was 7 days.

Two theses have shown that these recommendations were poorly applied in geriatric services. Indeed, the duration of treatment exceeded 7 days, and less than 30% of antibiotic antibiotic treatments were re-evaluated at 72 hours.

In 2021, the SPLIF ( published new recommendations reducing this duration to 5 days in the event of clinical improvement observed on the 3rd day of treatment. These new recommendations are based on studies, in which the average age of participants was 65 years. However, the average age of patients in geriatric short-stay departments is 84.7 years.

In addition, the geriatric population is characterized by immunosenescence, pulmonary vulnerability and undernutrition, raising questions about the validity of these recommendations in the geriatric population.

The investigators offer a monocentric, retrospective, observational study of the geriatric hospital Casanova to assess the application of SPLIF recommendations in the geriatric population.

ELIGIBILITY:
Inclusion Criteria:

* All patient treated for bacterial/community/nosocomial pneumonia who stayed in the geriatric short-stay at Casanova's Hospital between January 2, 2023 and April 30, 2023

Exclusion Criteria:

* HIV Positif
* Immunosupressed patient
* Complicated pneumonia (abcess, pleuropneumonia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the geriatric short-stay unit at the Casanova's hospital in Seine-saint-Denis for pneumopathy, between January 2, 2023 and April 30, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Sex | Day 1
Age | Day 1
Weight | Day 1
Phone Number | Day 1
Origins | Day 1
  Coming from Home, An institution...
Autonomy in daily life's score before hospitalisation | Day 1
  score between 0 (autonomous) and 6 (dependent)
Charlson's morbidity score | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Louise BORIES, Principal Investigator — Hôpital Delafontaine
Locations (1):
- Centre Hopitalier de Saint-Denis, Saint-Denis, Seine Saint Denis, France